CLINICAL TRIAL: NCT01014442
Title: Pharmacokinetics of Mycophenolate Mofetil in de Novo Lung Allograft Recipients
Brief Title: A Study of Mycophenolate Mofetil (CellCept) in Lung Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22608; 2009-012231-15
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2015-07

CONDITIONS: Lung Transplantation
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- Mycophenolate Mofetil; Cystic Fibrosis (Experimental): Participants with cystic fibrosis will receive mycophenolate mofetil 1.5 g, orally (PO), BID from Days 2 through 30 post-transplantation, and 1 g, PO, BID from Days 31 through 90 post-transplantation.
  Interventions: Drug: mycophenolate mofetil
- Mycophenolate Mofetil; Other (Experimental): Participants with COPD, emphysema, idiopathic pulmonary fibrosis, or A1AD will receive mycophenolate mofetil 1.5 g, PO, BID, from Days 2 through 30 post-transplantation, and 1 g, PO, BID from Days 31 through 90 post-transplantation.
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — 1.5 g PO BID from Days 2 to 30 post-transplantation, 1 g PO BID Days 31 to 90 post-transplantation
  Other Names: CellCept

SUMMARY:
This open-label, single center study will assess the pharmacokinetics, efficacy and safety of mycophenolate mofetil in lung allograft recipients. Participants will be split into 2 groups according to the original disease: Group A (cystic fibrosis) and Group B (chronic obstructive pulmonary disease [COPD], emphysema, idiopathic pulmonary fibrosis, alpha-1 antitrypsin deficiency [A1AD]). All participants will receive mycophenolate mofetil orally, 1.5 grams (g) twice daily (BID) from Day 2 to 30 post transplantation, and 1 g BID from Day 31 to 90 post transplantation. Anticipated time on study treatment is 90 days, and target sample size is 50-100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* primary single or bilateral lung allograft
* original disease cystic fibrosis, COPD, emphysema, idiopathic pulmonary fibrosis or A1AD

Exclusion Criteria:

* lung allograft retransplantation
* multiple organ transplantation
* severe gastrointestinal disorder
* malignancies or history of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Department of Cardiothoracic, Transplantation and Vascular Surgery at Hannover Medical School, Hanover, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- MMF - Cystic Fibrosis: Participants with cystic fibrosis having transplantation at Day 0, received mycophenolate mofetil (MMF) capsules at dose of 1.5 grams (g) twice daily (BID) from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with chronic obstructive pulmonary disorder (COPD), emphysema, idiopathic pulmonary fibrosis (IPF), or alpha-1 antitrypsin deficiency (A1AD) having transplantation at Day 0, received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
Period: Overall Study
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Started | 33 | 35
Completed | 26 | 16
Not Completed | 7 | 19
Not completed — Adverse Event | 0 | 8
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Protocol Violation | 2 | 5
Not completed — Lack of Compliance | 0 | 1
Not completed — Unspecified Reason | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of study drug and a safety follow-up, whether withdrawn prematurely or not.
Groups:
- MMF - Cystic Fibrosis: Participants with cystic fibrosis having transplantation at Day 0, received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD having transplantation at Day 0, received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
- Total: Total of all reporting groups
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.42) | 54.3 (7.93) | 43.1 (13.86)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Mycophenolic Acid (MPA), Mycophenolic Acid Glucuronide (MPAG) and Acyl Glucuronide Metabolite of Mycophenolic Acid (AcMPAG) at Day 4
Description: Cmax was expressed in milligrams per liter (mg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 after transplantation
Population: Per Protocol (PP) Population: Intent-to treat (ITT) population (received at least one dose of study drug and where the primary variable was measured at least once under study drug) excluding participants with major protocol violations (total 46 participants). Number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
mg/L
  MPA | 7.914 (5.46450) | 5.608 (2.5591)
  MPAG | 117.210 (58.9632) | 91.207 (26.3876)
  AcMPAG | 1.583 (0.9697) | 1.810 (0.8306)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2649, Wilcoxon rank sum test; Hodges-Lehmann estimator = 1.305, 95% CI 2-sided [-0.8300 to 4.2500]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3113, Wilcoxon rank sum test; Hodges-Lehmann estimator = 11.405, 95% CI 2-sided [-10.2000 to 42.7800]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2953, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.305, 95% CI 2-sided [-0.8100 to 0.1900]

2. Primary Outcome: Cmax of MPA, MPAG and AcMPAG at Day 8
Description: Cmax was expressed in mg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD, received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
mg/L
  MPA | 5.124 (4.2748) | 6.106 (3.3663)
  MPAG | 100.127 (54.0215) | 100.128 (25.1228)
  AcMPAG | 1.007 (0.5914) | 1.361 (0.9163)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1308, Wilcoxon rank sum test; Hodges-Lehmann estimator = -1.29, 95% CI 2-sided [-2.9900 to 0.4100]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4886, Wilcoxon rank sum test; Hodges-Lehmann estimator = -10.845, 95% CI 2-sided [-31.5000 to 20.7900]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2218, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.2, 95% CI 2-sided [-0.6000 to 0.1900]

3. Primary Outcome: Cmax of MPA, MPAG and AcMPAG at Day 20
Description: Cmax was expressed in mg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD, having transplantation at Day 0 received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
mg/L
  MPA | 5.284 (3.8472) | 6.762 (3.7405)
  MPAG | 93.882 (37.6112) | 124.450 (45.0613)
  AcMPAG | 0.624 (0.3895) | 1.434 (1.0501)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0886, Wilcoxon rank sum test; Hodges-Lehmann estimator = -1.87, 95% CI 2-sided [-3.7900 to 0.2800]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0220, Wilcoxon rank sum test; Hodges-Lehmann estimator = -30.76, 95% CI 2-sided [-54.9700 to -6.3600]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0008, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.56, 95% CI 2-sided [-1.0200 to -0.2700]

4. Primary Outcome: Cmax of MPA, MPAG and AcMPAG at Day 90
Description: Cmax was expressed in mg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
mg/L
  MPA | 12.915 (9.2479) | 7.294 (3.1817)
  MPAG | 104.938 (44.6135) | 113.453 (48.2935)
  AcMPAG | 1.375 (0.6514) | 1.163 (0.6856)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0318, Wilcoxon rank sum test; Hodges-Lehmann estimator = 3.945, 95% CI 2-sided [0.2500 to 8.2300]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.7144, Wilcoxon rank sum test; Hodges-Lehmann estimator = -7.59, 95% CI 2-sided [-51.1900 to 30.7000]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of AcMPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3930, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.27, 95% CI 2-sided [-0.3100 to 0.8800]

5. Primary Outcome: Cmax of Free MPA at Day 4
Description: Cmax was expressed in micrograms per liter (mcg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 23
mcg/L | 135.275 (133.2231) | 84.014 (57.8348)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of Free MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3002, Wilcoxon rank sum test; Hodges-Lehmann estimator = 17.08, 95% CI 2-sided [-16.5000 to 74.3200]

6. Primary Outcome: Cmax of Free MPA at Day 8
Description: Cmax was expressed in mcg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 18 | 21
mcg/L | 59.571 (35.1104) | 95.553 (62.6051)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of Free MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0334, Wilcoxon rank sum test; Hodges-Lehmann estimator = -25.24, 95% CI 2-sided [-53.2500 to -2.2900]

7. Primary Outcome: Cmax of Free MPA at Day 20
Description: Cmax was expressed in mcg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 16 | 20
mcg/L | 51.822 (39.9533) | 100.094 (120.8269)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of Free MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1151, Wilcoxon rank sum test; Hodges-Lehmann estimator = -23.805, 95% CI 2-sided [-52.2700 to 5.9700]

8. Primary Outcome: Cmax of Free MPA at Day 90
Description: Cmax was expressed in mcg/L.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 11 | 10
mcg/L | 87.293 (97.6509) | 101.472 (93.9834)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmax of Free MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.5974, Wilcoxon rank sum test; Hodges-Lehmann estimator = -15.63, 95% CI 2-sided [-63.8800 to 30.5600]

9. Primary Outcome: Dose-Normalized Cmax of MPA, MPAG, AcMPAG and Free MPA at Day 4
Description: Dose-normalized Cmax was determined (in 1 per liter [1/L]) by dividing the Cmax by the actual dose taken.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure. Number of participants with available data for specified category are provided against individual category.
Measure: Mean (Standard Deviation); unit: 1/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
1/L
  MPA | 0.00557 (0.003907) | 0.00422 (0.001924)
  MPAG | 0.08286 (0.037461) | 0.06749 (0.017478)
  AcMPAG | 0.001122 (0.0006350) | 0.001388 (0.0007160)
  Free MPA: number analyzed (Participants) | 19 | 23
  Free MPA | 0.0000929 (0.00008796) | 0.0000625 (0.00003907)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.5466, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0005, 95% CI 2-sided [-0.00103 to 0.00259]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3223, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.00728, 95% CI 2-sided [-0.00707 to 0.03161]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2108, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00026, 95% CI 2-sided [-0.00070 to 0.00012]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of Free MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called a Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4334, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0000112, 95% CI 2-sided [-0.0000140 to 0.0000462]

10. Primary Outcome: Dose-Normalized Cmax of MPA, MPAG, AcMPAG and Free MPA at Day 8
Description: Dose-normalized Cmax was determined (in 1/L) by dividing the Cmax by the actual dose taken.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
1/L
  MPA | 0.00356 (0.002769) | 0.00435 (0.002522)
  MPAG | 0.06980 (0.033524) | 0.07070 (0.017856)
  AcMPA | 0.000702 (0.0003736) | 0.000967 (0.0006297)
  Free MPA: number analyzed (Participants) | 18 | 21
  Free MPA | 0.0000409 (0.00002274) | 0.0000663 (0.00004075)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1511, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00081, 95% CI 2-sided [-0.00216 to 0.00030]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4131, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00695, 95% CI 2-sided [-0.02050 to 0.01103]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2677, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00017, 95% CI 2-sided [-0.00046 to 0.00013]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of Free MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0173, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0000185, 95% CI 2-sided [-0.0000394 to -0.0000050]

11. Primary Outcome: Dose-Normalized Cmax of MPA, MPAG, AcMPAG and Free MPA at Day 20
Description: Dose-normalized Cmax was determined (in 1/L) by dividing the Cmax by the actual dose taken.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
1/L
  MPA | 0.00395 (0.002619) | 0.00456 (0.002462)
  MPAG | 0.07044 (0.029284) | 0.08430 (0.029430)
  AcMPAG | 0.000482 (0.0003487) | 0.000969 (0.0006947)
  Free MP: number analyzed (Participants) | 16 | 20
  Free MP | 0.0000439 (0.00004750) | 0.0000666 (0.00008052)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis; Dose-Normalized Cmax of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3784, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00063, 95% CI 2-sided [-0.00230 to 0.00084]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0942, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.01602, 95% CI 2-sided [-0.03229 to 0.00297]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0032, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00037, 95% CI 2-sided [-0.00062 to -0.00015]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of Free MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1760, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0000126, 95% CI 2-sided [-0.0000328 to -0.0000091]

12. Primary Outcome: Dose-Normalized Cmax of MPA, MPAG, AcMPAG and Free MPA at Day 90
Description: Dose-normalized Cmax was determined (in 1/L) by dividing the Cmax by the actual dose taken.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 16 | 12
1/L
  MPA: number analyzed (Participants) | 15 | 12
  MPA | 0.01261 (0.007644) | 0.00742 (0.003631)
  MPAG: number analyzed (Participants) | 15 | 12
  MPAG | 0.10671 (0.037035) | 0.10948 (0.030395)
  AcMPAG | 0.001377 (0.0006935) | 0.001134 (0.0005100)
  Free MPA: number analyzed (Participants) | 11 | 10
  Free MPA | 0.0000945 (0.00009640) | 0.0001043 (0.00009208)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0509, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0043, 95% CI 2-sided [-0.00027 to 0.00833]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8262, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00567, 95% CI 2-sided [-0.03414 to 0.02671]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4345, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.00023, 95% CI 2-sided [-0.00030 to 0.00070]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized Cmax of Free MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.6472, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00001, 95% CI 2-sided [-0.0000586 to 0.0000364]

13. Primary Outcome: Time to Maximum Concentration (Tmax) of MPA, MPAG, AcMPAG and Free MPA at Day 4
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
hour
  MPA | 1.823 (1.1626) | 2.892 (2.9202)
  MPAG | 3.713 (2.4167) | 4.891 (2.6546)
  AcMPAG | 2.379 (1.2344) | 3.405 (1.9162)
  Free MPA: number analyzed (Participants) | 19 | 23
  Free MPA | 1.472 (0.3758) | 1.405 (0.4644)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.5745, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0333, 95% CI 2-sided [-1.9500 to 0.5000]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2003, Wilcoxon rank sum test; Hodges-Lehmann estimator = -1.8, 95% CI 2-sided [-2.3333 to 0.0833]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of AcMPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0929, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.5, 95% CI 2-sided [-2.0833 to 0.0000]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of Free MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0823, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0, 95% CI 2-sided [0.0000 to 0.0667]

14. Primary Outcome: Tmax of MPA, MPAG, AcMPAG and Free MPA at Day 8
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
hour
  MPA | 2.138 (1.4976) | 1.659 (0.9530)
  MPAG | 3.669 (1.4773) | 3.647 (1.4555)
  AcMPAG | 2.802 (1.2418) | 2.546 (1.1508)
  Free MPA: number analyzed (Participants) | 18 | 21
  Free MPA | 1.272 (0.5982) | 1.446 (0.3638)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8106, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0417, 95% CI 2-sided [-0.5000 to 1.7333]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 1.0000, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0, 95% CI 2-sided [-0.1667 to 0.1667]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.6311, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0667, 95% CI 2-sided [-0.3333 to 1.4667]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of Free MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4330, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0, 95% CI 2-sided [-0.1667 to 0.0167]

15. Primary Outcome: Tmax of MPA, MPAG, AcMPAG and Free MPA at Day 20
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
hour
  MPA | 2.293 (1.9048) | 2.463 (1.8928)
  MPAG | 3.762 (2.2954) | 4.907 (2.8568)
  AcMPAG | 2.842 (1.7915) | 3.411 (1.8799)
  Free MPA: number analyzed (Participants) | 16 | 20
  Free MPA | 1.236 (0.6144) | 1.366 (0.4692)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 1.0000, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0, 95% CI 2-sided [-1.1667 to 0.5833]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4947, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0833, 95% CI 2-sided [-2.0000 to 0.0833]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4425, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.1667, 95% CI 2-sided [-1.9667 to 0.2000]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of Free MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9720, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0, 95% CI 2-sided [-0.0500 to 0.0333]

16. Primary Outcome: Tmax of MPA, MPAG, AcMPAG and Free MPA at Day 90
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
hour
  MPA | 1.450 (0.5251) | 2.143 (2.2487)
  MPAG | 3.095 (1.7884) | 4.420 (1.9078)
  AcMPAG | 2.234 (1.0899) | 3.564 (2.3686)
  Free MPA: number analyzed (Participants) | 11 | 10
  Free MPA | 1.490 (0.0666) | 1.485 (0.5282)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8834, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0333, 95% CI 2-sided [-1.1667 to 0.7000]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0386, Wilcoxon rank sum test; Hodges-Lehmann estimator = -1.8333, 95% CI 2-sided [-2.2000 to 0.0000]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0558, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.525, 95% CI 2-sided [-2.6167 to 0.0000]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Tmax of Free MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0082, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.15, 95% CI 2-sided [-0.2333 to -0.0667]

17. Primary Outcome: Minimum Concentration (Cmin) of MPA, MPAG and AcMPAG at Day 4
Description: Cmin was expressed in mg/L.
Time Frame: Predose (0 hour) on Day 4 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 25
mg/L
  MPA | 1.267 (1.0082) | 1.094 (0.8473)
  MPAG | 66.917 (41.3384) | 47.493 (17.9747)
  AcMPAG: number analyzed (Participants) | 21 | 24
  AcMPAG | 0.602 (0.5628) | 0.733 (0.4686)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.5224, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.13, 95% CI 2-sided [-0.2600 to 0.5000]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2088, Wilcoxon rank sum test; Hodges-Lehmann estimator = 11.16, 95% CI 2-sided [-5.2900 to 30.2900]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1794, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.165, 95% CI 2-sided [-0.4500 to 0.0800]

18. Primary Outcome: Cmin of MPA, MPAG and AcMPAG at Day 8
Description: Cmin was expressed in mg/L.
Time Frame: Predose (0 hour) on Day 8 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 24
mg/L
  MPA | 0.750 (0.6136) | 0.772 (0.3482)
  MPAG | 54.566 (51.2379) | 57.189 (20.8518)
  AcMPAG: number analyzed (Participants) | 17 | 22
  AcMPAG | 0.386 (0.4870) | 0.517 (0.2623)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4027, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.125, 95% CI 2-sided [-0.3800 to 0.1900]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0875, Wilcoxon rank sum test; Hodges-Lehmann estimator = -16.09, 95% CI 2-sided [-29.3500 to 6.3900]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0112, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.2, 95% CI 2-sided [-0.3500 to -0.0500]

19. Primary Outcome: Cmin of MPA, MPAG and AcMPAG at Day 20
Description: Cmin was expressed in mg/L.
Time Frame: Predose (0 hour) on Day 20 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 18 | 22
mg/L
  MPA | 0.782 (0.5945) | 1.234 (0.9971)
  MPAG | 58.484 (29.5576) | 69.023 (25.6603)
  AcMPAG: number analyzed (Participants) | 13 | 22
  AcMPAG | 0.261 (0.1662) | 0.528 (0.3977)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0818, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.215, 95% CI 2-sided [-0.5600 to 0.0500]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0945, Wilcoxon rank sum test; Hodges-Lehmann estimator = -14.03, 95% CI 2-sided [-26.9000 to 2.9400]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0081, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.19, 95% CI 2-sided [-0.4100 to -0.0400]

20. Primary Outcome: Cmin of MPA, MPAG and AcMPAG at Day 90
Description: Cmin was expressed in mg/L.
Time Frame: Predose (0 hour) on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
mg/L
  MPA | 1.103 (0.7446) | 1.570 (1.0282)
  MPAG | 57.957 (32.6863) | 80.488 (37.2631)
  AcMPAG: number analyzed (Participants) | 13 | 12
  AcMPAG | 0.449 (0.3552) | 0.466 (0.3096)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3289, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.36, 95% CI 2-sided [-1.1400 to 0.2800]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1243, Wilcoxon rank sum test; Hodges-Lehmann estimator = -20.3, 95% CI 2-sided [-49.3900 to 4.7100]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Cmin of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8704, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.03, 95% CI 2-sided [-0.2800 to 0.2300]

21. Primary Outcome: Cmin of Free MPA at Day 4
Description: Cmin was expressed in mcg/L.
Time Frame: Predose (0 hour) on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 23
mcg/L | 40.188 (37.9357) | 23.711 (14.6991)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4043, Wilcoxon rank sum test; Hodges-Lehmann estimator = 5.22, 95% CI 2-sided [-5.0100 to 24.4900]

22. Primary Outcome: Cmin of Free MPA at Day 8
Description: Cmin was expressed in mcg/L.
Time Frame: Predose (0 hour) on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Groups:
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD, having transplantation at Day 0 received MMF at dose of 1.5 g BID from Day 2 to Day 30 post-transplantation and then at 1 g BID from Day 31 to Day 90 post-transplantation.
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 24
mcg/L | 18.161 (16.3831) | 15.669 (9.6168)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.8930, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.44, 95% CI 2-sided [-6.0700 to 8.0100]

23. Primary Outcome: Cmin of Free MPA at Day 20
Description: Cmin was expressed in mcg/L.
Time Frame: Predose (0 hour) on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 18 | 20
mcg/L | 12.193 (9.1443) | 20.237 (16.2117)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.0819, Wilcoxon rank sum test; Hodges-Lehmann estimator = -4.935, 95% CI 2-sided [-14.3100 to 1.1100]

24. Primary Outcome: Cmin of Free MPA at Day 90
Description: Cmin was expressed in mcg/L.
Time Frame: Predose (0 hour) on Day 90 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 13 | 12
mcg/L | 8.102 (3.3201) | 18.831 (12.6155)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.0414, Wilcoxon rank sum test; Hodges-Lehmann estimator = -8.205, 95% CI 2-sided [-19.2700 to -0.0700]

25. Primary Outcome: Volume of Distribution (Vz) of MPA, MPAG and AcMPAG at Day 4
Description: Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 23
Liter
  MPA: number analyzed (Participants) | 21 | 22
  MPA | 345.46 (182.247) | 287.74 (237.295)
  MPAG: number analyzed (Participants) | 20 | 22
  MPAG | 11.681 (4.7587) | 12.062 (3.7316)
  AcMPAG: number analyzed (Participants) | 20 | 23
  AcMPAG | 1065.02 (611.137) | 705.38 (502.996)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1552, Wilcoxon rank sum test; Hodges-Lehmann estimator = 69.7186, 95% CI 2-sided [-23.4659 to 162.9545]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.6057, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.7836, 95% CI 2-sided [-3.2675 to 2.5529]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0188, Wilcoxon rank sum test; Hodges-Lehmann estimator = 299.1021, 95% CI 2-sided [79.5869 to 695.1789]

26. Primary Outcome: Vz of MPA, MPAG and AcMPAG at Day 8
Description: as for outcome 25
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 21
Liter
  MPA | 465.45 (260.837) | 331.51 (150.037)
  MPAG | 12.168 (5.1048) | 12.740 (5.2593)
  AcMPAG: number analyzed (Participants) | 19 | 20
  AcMPAG | 1432.88 (919.423) | 1173.38 (708.767)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0659, Wilcoxon rank sum test; Hodges-Lehmann estimator = 88.959, 95% CI 2-sided [-5.7876 to 209.0183]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.7842, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.4456, 95% CI 2-sided [-3.1366 to 2.2920]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4072, Wilcoxon rank sum test; Hodges-Lehmann estimator = 121.3737, 95% CI 2-sided [-233.6483 to 560.0069]

27. Primary Outcome: Vz of MPA, MPAG and AcMPAG at Day 20
Description: as for outcome 25
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
Liter
  MPA | 476.06 (267.025) | 257.57 (126.679)
  MPAG: number analyzed (Participants) | 16 | 17
  MPAG | 12.798 (5.1535) | 9.533 (3.1984)
  AcMPAG: number analyzed (Participants) | 13 | 21
  AcMPAG | 3006.18 (2570.205) | 1571.93 (1944.621)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0040, Wilcoxon rank sum test; Hodges-Lehmann estimator = 207.9933, 95% CI 2-sided [71.2442 to 355.1739]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0689, Wilcoxon rank sum test; Hodges-Lehmann estimator = 2.6186, 95% CI 2-sided [-0.1999 to 6.7766]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0306, Wilcoxon rank sum test; Hodges-Lehmann estimator = 635.7812, 95% CI 2-sided [49.4696 to 2793.7642]

28. Primary Outcome: Vz of MPA, MPAG and AcMPAG at Day 90
Description: as for outcome 25
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
Liter
  MPA | 139.48 (78.679) | 192.53 (226.826)
  MPAG: number analyzed (Participants) | 12 | 8
  MPAG | 9.254 (4.6738) | 9.201 (4.4274)
  AcMPAG: number analyzed (Participants) | 12 | 9
  AcMPAG | 811.15 (404.733) | 980.49 (473.444)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9029, Wilcoxon rank sum test; Hodges-Lehmann estimator = 4.7477, 95% CI 2-sided [-73.5212 to 59.8304]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9692, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0077, 95% CI 2-sided [-3.6739 to 3.9521]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Vz of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3744, Wilcoxon rank sum test; Hodges-Lehmann estimator = -149.7962, 95% CI 2-sided [-644.4526 to 311.9735]

29. Primary Outcome: Clearance (CL) of MPA, MPAG and AcMPAG at Day 4
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body and expressed in liters per hour (L/hour).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: L/hours
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
L/hours
  MPA | 68.471 (32.7611) | 56.709 (22.3503)
  MPAG | 1.6754 (0.81910) | 1.7615 (0.46573)
  AcMPAG | 206.60 (151.301) | 140.96 (110.400)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1362, Wilcoxon rank sum test; Hodges-Lehmann estimator = 7.8422, 95% CI 2-sided [-3.9110 to 18.4444]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4325, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.1609, 95% CI 2-sided [-0.5693 to 0.2710]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0316, Wilcoxon rank sum test; Hodges-Lehmann estimator = 47.2686, 95% CI 2-sided [4.1970 to 112.7806]

30. Primary Outcome: CL of MPA, MPAG and AcMPAG at Day 8
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body and expressed in L/hour.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
L/hour
  MPA | 90.921 (33.7184) | 81.578 (63.7936)
  MPAG | 2.3235 (1.55336) | 1.7847 (0.75624)
  AcMPAG | 410.86 (448.947) | 253.81 (237.283)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0572, Wilcoxon rank sum test; Hodges-Lehmann estmator = 19.0536, 95% CI 2-sided [-0.4250 to 35.3852]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3198, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.3541, 95% CI 2-sided [-0.2524 to 1.1097]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0845, Wilcoxon rank sum test; Hodges-Lehmann estimator = 54.0322, 95% CI 2-sided [-6.7706 to 160.3469]

31. Primary Outcome: CL of MPA, MPAG and AcMPAG at Day 20
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body and expressed in L/hour.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
L/hour
  MPA | 83.068 (27.7321) | 58.295 (19.5800)
  MPAG | 1.9338 (0.69979) | 1.4788 (0.44488)
  AcMPAG | 680.68 (614.970) | 232.34 (179.449)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0048, Wilcoxon rank sum test; Hodges-Lehmann estimator = 25.0037, 95% CI 2-sided [8.2373 to 43.5102]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0277, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.4297, 95% CI 2-sided [0.0340 to 0.9925]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0002, Wilcoxon rank sum test; Hodges-Lehmann estimator = 318.5455, 95% CI 2-sided [154.1902 to 526.1716]

32. Primary Outcome: CL of MPA, MPAG and AcMPAG at Day 90
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body and expressed in L/hour.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
L/hour
  MPA | 38.091 (20.9125) | 36.922 (15.2129)
  MPAG | 1.5701 (0.99265) | 1.2433 (0.53337)
  AcMPAG: number analyzed (Participants) | 14 | 12
  AcMPAG | 231.28 (218.455) | 223.56 (191.887)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9417, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.579, 95% CI 2-sided [-14.5052 to 11.6346]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2941, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.1817, 95% CI 2-sided [-0.1954 to 0.6246]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; CL of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8170, Wilcoxon rank sum test; Hodges-Lehmann estimator = -4.9076, 95% CI 2-sided [-84.8234 to 109.9321]

33. Primary Outcome: Area Under the Curve From Time 0 to 12 Hours (AUC0-12) of MPA, MPAG and AcMPAG at Day 4
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours time milligrams per liter (hours*[mg/L]).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*(mg/L)
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
hours*(mg/L)
  MPA | 23.460 (7.8103) | 27.174 (10.4909)
  MPAG | 1095.98 (659.211) | 829.14 (281.878)
  AcMPAG | 10.414 (7.5535) | 13.672 (6.6349)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2798, Wilcoxon rank sum test; Hodges-Lehmann estimator = -2.4102, 95% CI 2-sided [-8.5642 to 3.0044]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4063, Wilcoxon rank sum test; Hodges-Lehmann estimator = 72.7203, 95% CI 2-sided [-107.1596 to 393.5295]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0441, Wilcoxon rank sum test; Hodges-Lehmann estimator = -3.6042, 95% CI 2-sided [-8.1854 to -0.1887]

34. Primary Outcome: AUC0-12 of MPA, MPAG and AcMPAG at Day 8
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*(mg/L)
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
hours*(mg/L)
  MPA | 17.841 (8.2077) | 23.352 (10.7853)
  MPAG | 881.50 (634.587) | 888.96 (277.565)
  AcMPAG | 6.064 (4.2591) | 9.081 (6.5063)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0510, Wilcoxon rank sum test; Hodges-Lehmann estimator = -5.8077, 95% CI 2-sided [-11.7302 to 0.0033]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2733, Wilcoxon rank sum test; Hodges-Lehmann estimator = -171.159, 95% CI 2-sided [-361.4437 to 171.9652]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0718, Wilcoxon rank sum test; Hodges-Lehmann estimator = -1.9621, 95% CI 2-sided [-4.8456 to 0.2067]

35. Primary Outcome: AUC0-12 of MPA, MPAG and AcMPAG at Day 20
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*(mg/L)
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
hours*(mg/L)
  MPA | 18.925 (10.7674) | 28.290 (10.5485)
  MPAG | 812.65 (391.881) | 1095.37 (391.620)
  AcMPAG | 3.252 (2.2066) | 9.482 (6.6815)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0002, Wilcoxon rank sum test; Hodges-Lehmann estimator = -8.6964, 95% CI 2-sided [-13.7713 to -4.6498]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0058, Wilcoxon rank sum test; Hodges-Lehmann estimator = -268.9537, 95% CI 2-sided [-506.7782 to -77.3970]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test; Hodges-Lehmann estimator = -4.828, 95% CI 2-sided [-7.1455 to -2.6133]

36. Primary Outcome: AUC0-12 of MPA, MPAG and AcMPAG at Day 90
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours*(mg/L)
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
hours*(mg/L)
  MPA | 32.365 (16.4658) | 31.864 (15.5442)
  MPAG | 776.28 (385.310) | 972.69 (530.667)
  AcMPAG: number analyzed (Participants) | 14 | 12
  AcMPAG | 7.776 (5.0791) | 7.219 (5.2217)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.7144, Wilcoxon rank sum test; Hodges-Lehmann estimator = 1.7477, 95% CI 2-sided [-12.1010 to 14.6563]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3413, Wilcoxon rank sum test; Hodges-Lehmann estimator = -156.3255, 95% CI 2-sided [-526.0765 to 195.8348]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; AUC0-12 of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.6251, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.888, 95% CI 2-sided [-3.0288 to 4.2273]

37. Primary Outcome: AUC0-12 of Free MPA at Day 4
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours times micrograms per liter (hours*[mcg/L]).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 22
hours*mcg/L | 135.703 (120.4152) | 80.272 (45.9523)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.2342, Wilcoxon rank sum test; Hodges-Lehmann estimator = 24.315, 95% CI 2-sided [-16.0292 to 79.3650]

38. Primary Outcome: AUC0-12 of Free MPA at Day 8
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mcg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
hours*mcg/L | 61.155 (26.0913) | 83.683 (51.4228)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.1964, Wilcoxon rank sum test; Hodges-Lehmann estimator = -13.5592, 95% CI 2-sided [-37.3950 to 5.4825]

39. Primary Outcome: AUC0-12 of Free MPA at Day 20
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mcg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 16 | 20
hours*mcg/L | 48.530 (30.3408) | 89.315 (90.3819)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.0672, Wilcoxon rank sum test; Hodges-Lehmann estimator = -22.7878, 95% CI 2-sided [-44.8217 to 3.7573]

40. Primary Outcome: AUC0-12 of Free MPA at Day 90
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours and expressed in hours*(mcg/L).
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mcg/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 11 | 10
hours*mcg/L | 68.874 (64.6536) | 99.212 (81.0812)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.2453, Wilcoxon rank sum test; Hodges-Lehmann estimator = -21.4737, 95% CI 2-sided [-64.1567 to 8.5708]

41. Primary Outcome: Dose-Normalized AUC0-12 of MPA, MPAG, AcMPAG and Free MPA at Day 4
Description: AUC0-12 is a measure of the serum concentration of the drug from time 0 to 12 hours. Dose-normalized AUC0-12 was determined (in hours/L) by dividing the AUC0-12 by the actual dose taken.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 21 | 24
hours/L
  MPA | 0.01652 (0.004684) | 0.02016 (0.007383)
  MPAG | 0.7720 (0.42519) | 0.6165 (0.20281)
  AcMPAG | 0.00739 (0.005002) | 0.01056 (0.005828)
  Free MPA: number analyzed (Participants) | 19 | 22
  Free MPA | 0.0000943 (0.00008029) | 0.0000594 (0.00003237)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1362, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00237, 95% CI 2-sided [-0.00734 to 0.00106]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 MPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.4325, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.04797, 95% CI 2-sided [-0.08467 to 0.26322]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of AcMPAG at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0316, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00311, 95% CI 2-sided [-0.00645 to -0.00029]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of Free MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3269, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0000158, 95% CI 2-sided [-0.0000134 to 0.0000552]

42. Primary Outcome: Dose-Normalized AUC0-12 of MPA, MPAG, AcMPAG and Free MPA at Day 8
Description: as for outcome 41
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 22
hours/L
  MPA | 0.01256 (0.005018) | 0.01624 (0.007077)
  MPAG | 0.6157 (0.40835) | 0.6270 (0.18884)
  AcMPAG | 0.00426 (0.002733) | 0.00644 (0.004471)
  Free MPA: number analyzed (Participants) | 17 | 21
  Free MPA | 0.0000428 (0.00001807) | 0.0000580 (0.00003330)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0572, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00383, 95% CI 2-sided [-0.00761 to 0.00010]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3198, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.09626, 95% CI 2-sided [-0.25269 to 0.11464]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of AcMPAG at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0845, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00131, 95% CI 2-sided [-0.00352 to 0.00013]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of Free MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1769, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.00001, 95% CI 2-sided [-0.0000250 to 0.0000043]

43. Primary Outcome: Dose-Normalized AUC0-12 of MPA, MPAG, AcMPAG and Free MPA at Day 20
Description: as for outcome 41
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
hours/L
  MPA | 0.01402 (0.007208) | 0.01923 (0.007029)
  MPAG | 0.6059 (0.28149) | 0.7440 (0.26032)
  AcMPAG | 0.00239 (0.001707) | 0.00642 (0.004432)
  Free MPA: number analyzed (Participants) | 16 | 20
  Free MPA | 0.0000399 (0.00003632) | 0.0000597 (0.00006020)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0048, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0049, 95% CI 2-sided [-0.00876 to -0.00148]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0277, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.14764, 95% CI 2-sided [-0.31026 to -0.01067]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of AcMPAG at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0002, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0035, 95% CI 2-sided [-0.00476 to 0.00168]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of Free MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1661, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0000138, 95% CI 2-sided [-0.0000295 to 0.0000047]

44. Primary Outcome: Dose-Normalized AUC0-12 of MPA, MPAG, AcMPAG and Free MPA at Day 90
Description: as for outcome 41
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours/L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 15 | 12
hours/L
  MPA | 0.03126 (0.011529) | 0.03172 (0.012879)
  MPAG | 0.7887 (0.31007) | 0.9190 (0.31896)
  AcMPAG: number analyzed (Participants) | 14 | 12
  AcMPAG | 0.00748 (0.004735) | 0.00700 (0.004084)
  Free MPA: number analyzed (Participants) | 11 | 10
  Free MPA | 0.0000752 (0.00006364) | 0.00001023 (0.00007888)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9417, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.00054, 95% CI 2-sided [-0.01037 to 0.01042]
Statistical Analysis 2: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of MPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2941, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.1461, 95% CI 2-sided [-0.39951 to 0.12988]
Statistical Analysis 3: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of AcMPAG at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.8170, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.00033, 95% CI 2-sided [-0.00361 to 0.00421]
Statistical Analysis 4: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Dose-Normalized AUC0-12 of Free MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.1927, Wilcoxon rank sum test; Hodge-Lehmann estimator = -0.0000239, 95% CI 2-sided [-0.0000594 to 0.0000154]

45. Primary Outcome: Free Fraction of Free MPA at Day 4
Description: MPA Free fraction (in percent [%]) was calculated by dividing free MPA AUC0-12 by total MPA AUC0-12 times 100%.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 4 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of free fraction
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 22
percentage of free fraction | 0.5789 (0.42113) | 0.3208 (0.16486)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Free Fraction of Free MPA at Day 4. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0821, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.1616, 95% CI 2-sided [-0.0121 to 0.4188]

46. Primary Outcome: Free Fraction of Free MPA at Day 8
Description: MPA Free fraction (in %) was calculated by dividing free MPA AUC0-12 by total MPA AUC0-12 times 100%.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 8 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of free fraction
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 17 | 21
percentage of free fraction | 0.3595 (0.13517) | 0.3594 (0.20504)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Free Fraction of Free MPA at Day 8. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.3628, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0427, 95% CI 2-sided [-0.0455 to 0.1221]

47. Primary Outcome: Free Fraction of Free MPA at Day 20
Description: MPA Free fraction (in %) was calculated by dividing free MPA AUC0-12 by total MPA AUC0-12 times 100%.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 20 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of free fraction
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 16 | 20
percentage of free fraction | 0.2922 (0.19811) | 0.3052 (0.22218)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Free Fraction of Free MPA at Day 20. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.9873, Wilcoxon rank sum test; Hodges-Lehmann estimator = 0.0010, 95% CI 2-sided [-0.1152 to 0.1173]

48. Primary Outcome: Free Fraction of Free MPA at Day 90
Description: MPA Free fraction (in %) was calculated by dividing free MPA AUC0-12 by total MPA AUC0-12 times 100%.
Time Frame: Predose (0 hour), 0.5, 1, 1.5, 2, 4, 8, 10, and 12 hours post-dose on Day 90 post-transplantation
Population: PP Population. Here, number of participants analyzed=participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of free fraction
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 11 | 10
percentage of free fraction | 0.2270 (0.14614) | 0.3020 (0.13446)
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Free Fraction of Free MPA at Day 90. Analysis was performed using Wilcoxon rank sum test; corresponding p-value and point estimate (Hodges-Lehmann estimator) were calculated. The point estimator derived by sending the confidence level to zero is called as Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.2178, Wilcoxon rank sum test; Hodges-Lehmann estimator = -0.0857, 95% CI 2-sided [-0.1870 to 0.0265]

49. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at Day 90 Post-Transplantation
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Day 90 post-transplantation
Population: ITT Population (total 64 participants). Here, Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 26 | 16
L | 3.087 (0.9335) | 2.834 (0.6912)

50. Secondary Outcome: Percent of Predicted FEV1 at Day 90 Post-Transplantation
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Percent predicted FEV1 [%] = (FEV1 [L] / Predicted normal value FEV1 [L]) * 100%
Time Frame: Day 90 post-transplantation
Population: ITT Population. Here, Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Groups:
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD, having transplantation at Day 0 received MMF at dose of 1.5 g BID from Day 2 to Day 30 and then at 1 g BID from Day 31 to Day 90.
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 26 | 15
percentage of predicted FEV1 | 81.75 (19.743) | 90.17 (20.176)

51. Secondary Outcome: Forced Vital Capacity (FVC) at Day 90 Post-Transplantation
Description: FVC at Day 90 post-transplantation is reported.
Time Frame: Day 90 post-transplantation
Population: ITT Population. Here, Number of participants analyzed = participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 26 | 16
L | 3.445 (0.9499) | 3.619 (1.0388)

52. Secondary Outcome: Change From Baseline in Intracellular Adenosine-Tri-Phosphate (iATP) Levels
Description: iATP was expressed in ng/mL.
Time Frame: Baseline, Days 4, 8, 20 and 90 post-transplantation
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome measure. Here "n"= participants who were evaluable for each category, for respective arm groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 20 | 18
ng/mL
  Day 4: number analyzed (Participants) | 19 | 18
  Day 4 | 24.0 (223.32) | 85.4 (215.78)
  Day 8: number analyzed (Participants) | 20 | 17
  Day 8 | 162.9 (294.53) | 144.9 (286.23)
  Day 20: number analyzed (Participants) | 15 | 15
  Day 20 | -42.4 (382.87) | -45.9 (199.20)
  Day 90: number analyzed (Participants) | 16 | 6
  Day 90 | -164.6 (312.98) | -114.7 (138.99)

53. Secondary Outcome: Change From Baseline in T-Cell Phenotype
Description: Reported values are change in the T-cell phenotype status from baseline to Day 20 and 90 for cluster of differentiation (CD) 3, CD19, CD4, CD4CD25, CD28, CD45RA, CD45RO, CD69, CD127, and CD152.
Time Frame: Baseline, Days 20 and 90 post-transplantation
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 19 | 16
percentage of lymphocytes
  CD3: Change at Day 20 | -1.34 (13.012) | -3.01 (13.075)
  CD3: Change at Day 90: number analyzed (Participants) | 11 | 8
  CD3: Change at Day 90 | 1.74 (11.433) | -2.81 (6.995)
  CD19: Change at Day 20 | 3.29 (10.554) | 1.88 (8.046)
  CD19: Change at Day 90: number analyzed (Participants) | 10 | 7
  CD19: Change at Day 90 | 0.59 (5.322) | 0.61 (6.000)
  CD4: Change at Day 20 | 13.29 (15.626) | -14.71 (24.467)
  CD4: Change at Day 90: number analyzed (Participants) | 10 | 8
  CD4: Change at Day 90 | 9.00 (26.054) | -1.93 (13.415)
  CD4CD25: Change at Day 20 | 2.72 (6.877) | -0.53 (0.940)
  CD4CD25: Change at Day 90: number analyzed (Participants) | 10 | 8
  CD4CD25: Change at Day 90 | 0.89 (1.354) | -0.10 (0.941)
  CD28: Change at Day 20: number analyzed (Participants) | 18 | 16
  CD28: Change at Day 20 | 4.54 (10.105) | -4.44 (7.635)
  CD28: Change at Day 90: number analyzed (Participants) | 10 | 8
  CD28: Change at Day 90 | 10.15 (25.362) | -1.04 (6.176)
  CD45RA: Change at Day 20 | 5.35 (15.802) | -5.11 (17.327)
  CD45RA: Change at Day 90: number analyzed (Participants) | 11 | 8
  CD45RA: Change at Day 90 | -1.57 (12.498) | -4.88 (13.342)
  CD45RO: Change at Day 20 | -0.08 (4.199) | -2.83 (3.285)
  CD45RO: Change at Day 90: number analyzed (Participants) | 12 | 8
  CD45RO: Change at Day 90 | -1.92 (7.564) | -0.43 (7.574)
  CD69: Change at Day 20 | 5.68 (10.031) | 0.01 (0.328)
  CD69: Change at Day 90: number analyzed (Participants) | 10 | 7
  CD69: Change at Day 90 | -0.46 (10.040) | -0.04 (0.237)
  CD127: Change at Day 20 | -1.36 (13.566) | -3.90 (7.227)
  CD127: Change at Day 90: number analyzed (Participants) | 10 | 7
  CD127: Change at Day 90 | -0.19 (14.603) | -2.03 (12.509)
  CD152: Change at Day 20 | -3.78 (17.562) | -10.97 (17.935)
  CD152: Change at Day 90: number analyzed (Participants) | 11 | 8
  CD152: Change at Day 90 | -0.28 (2.624) | -15.59 (29.715)

54. Secondary Outcome: Percentage of Participants With Opportunistic Infections
Description: Opportunistic infections included all infections which occurred due to aspergillus, candida, pneumocystis, cryptococcus, listeria, herpes zoster, herpes simplex, cytomegalovirus pathogens.
Time Frame: Up to Day 90
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Number analyzed (Participants) | 33 | 35
percentage of participants | 18.2 | 20.0
Statistical Analysis 1: Comparison: MMF - Cystic Fibrosis vs MMF - COPD, Emphysema, IPF, or A1AD; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Difference in rates = -1.8, 95% CI 2-sided [-24.9 to 22.1]

ADVERSE EVENTS:
Time Frame: From baseline up to Day 90
Groups:
- MMF - COPD, Emphysema, IPF, or A1AD: Participants with COPD, emphysema, IPF or A1AD, having transplantation at Day 0 received MMF capsules at dose of 1.5 g BID from Day 2 to Day 30 and then at 1 g BID from Day 31 to Day 90.
Arm/Group | MMF - Cystic Fibrosis | MMF - COPD, Emphysema, IPF, or A1AD
Serious Adverse Events (participants affected / at risk) | 13/33 | 14/35
Other Adverse Events (participants affected / at risk) | 27/33 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF - Cystic Fibrosis (N=33) | MMF - COPD, Emphysema, IPF, or A1AD (N=35)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Antibiotic resistant Staphylococcus test positive (Investigations) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumorthorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MMF - Cystic Fibrosis (N=33) | MMF - COPD, Emphysema, IPF, or A1AD (N=35)
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Hyperchromic anaemia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 3
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 12
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Visual impairment (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 4 | 4
Oedema peripheral (General disorders) | 0 | 3
Bacterial infection (Infections and infestations) | 3 | 4
Clostridium difficile colitis (Infections and infestations) | 3 | 0
Enterococcal infection (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 1 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 0 | 2
Pseudomonas infection (Infections and infestations) | 0 | 3
Anastomotic complication (Injury, poisoning and procedural complications) | 3 | 1
Antibody test positive (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 1 | 2
Klebsiella test positive (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 3 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Sleep disorder (Psychiatric disorders) | 0 | 6
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2 | 4
Circulatory collapse (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.